CLINICAL TRIAL: NCT02480582
Title: The Impact of Snacks Which Vary Nutritionally in Their Satiating Potential on Measures of Appetite Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Dr Graham Finlayson, Principal Investigator, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LDS-2015-ABC; RG.PSYC.102933 (Other Grant/Funding Number: Almond Board of California)
Record Dates: First submitted 2015-06-04; First posted 2015-06-24 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Lack of Satiety; Hyperphagia
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Almond, then No Food, then Cheese Savouries (Experimental): Participants first received a mid-morning snack of almonds (0.9g/kg). After a washout period of 5 days, they then received no food. Finally, after another washout period participants received a mid-morning snack of cheese savouries (0.9g/kg).
  Interventions: Other: Almonds; Other: Cheese Savouries
- Cheese Savouries then Almond, then No Food (Experimental): Participants first received a mid-morning snack of cheese savouries (0.9g/kg). After a washout period of 5 days, they then received a mid-morning snack of almonds (0.9g/kg). Finally, after another washout period participants received no food.
  Interventions: Other: Almonds; Other: Cheese Savouries
- No Food, then Cheese Savouries, then Almond (Experimental): Participants first received no food. After a washout period of 5 days, they then received a mid-morning snack of cheese savouries (0.9g/kg). Finally, after another washout period participants received a mid-morning snack of almonds (0.9g/kg).
  Interventions: Other: Almonds; Other: Cheese Savouries
- Cheese Savouries, then No Food, then Almond (Experimental): Participants first received a mid-morning snack of cheese savouries (0.9g\kg). After a washout period of 5 days, they then received no food. Finally, after another washout period participants received a mid-morning snack of almonds (0.9g\kg).
  Interventions: Other: Almonds; Other: Cheese Savouries
- Almond, then Cheese Savouries, then No Food (Experimental): Participants first received a mid-morning snack of almonds (0.9g\kg). After a washout period of 5 days, they then received a mid-morning snack of cheese savouries (0.9g\kg). Finally, after another washout period participants received no food.
  Interventions: Other: Almonds; Other: Cheese Savouries
- No Food, then Almond, then Cheese Savouries (Experimental): Participants first received no food. After a washout period of 5 days, they then received a mid-morning snack of almonds (0.9g/kg). Finally, after another washout period participants received a mid-morning snack of cheese savouries (0.9g\kg).
  Interventions: Other: Almonds; Other: Cheese Savouries

INTERVENTIONS:
Other: Almonds — Whole raw almonds provided as a mid-morning snack - 0.9g\kg
Other: Cheese Savouries — Cheese savoury crackers provided as a mid-morning snack - 0.9g/kg

SUMMARY:
The current study will examine the effect of almond consumption (0.9g/kg dose) compared to an energy and weight matched comparator food or no food on measures of appetite control including appetite sensations, energy intake and food hedonics.

DETAILED DESCRIPTION:
Some individuals exhibit a weak satiety response to food and may be susceptible to overconsumption. Snack foods can be substantial contributors to daily energy intake, with different types of snacks exerting potentially different effects on satiety per calorie consumed. The current study will compare the effect of consuming different snack foods on measures of appetite control including appetite sensations, energy intake and food hedonics in women with a weak satiety response.

In a crossover design, female participants will consume three different mid-morning snacks: raw almonds, savoury crackers or water. Appetite sensations, energy intake, food reward and craving will be assessed under controlled laboratory conditions. Satiety responsiveness will be determined using the satiety quotient (SQ).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided written informed consent.
* Healthy female participants aged 18-55 years.
* BMI of 18.5 - 30.0 kg/m2.
* Regular breakfast eaters.
* Not currently dieting to lose, gain or maintain weight.
* Non-smokers.
* Liking/acceptance of the study foods (≥4 on 7-point Likert scale).

Exclusion Criteria:

* Taking medication known to affect appetite within past month and/or during the study.
* Any known food allergies or food intolerances.
* Participants who do not regularly eat breakfast.
* Participants with low liking or acceptance of the study foods.
* Participants currently dieting to lose, gain or maintain weight.
* Reported history of or present eating disorder.
* BMI <18.5 kg/m2 or >30 kg/m2.
* Vegetarians.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Finlayson, PhD, Principal Investigator — University of Leeds

IPD SHARING:
Plan to Share IPD: Yes
Results to be written up for submission to peer-review scientific journal.

REFERENCES:
- [Background] Gibbons C, Caudwell P, Finlayson G, King N, Blundell J. Validation of a new hand-held electronic data capture method for continuous monitoring of subjective appetite sensations. Int J Behav Nutr Phys Act. 2011 Jun 8;8:57. doi: 10.1186/1479-5868-8-57. PMID 21651803
- [Background] Finlayson G, King N, Blundell J. The role of implicit wanting in relation to explicit liking and wanting for food: implications for appetite control. Appetite. 2008 Jan;50(1):120-7. doi: 10.1016/j.appet.2007.06.007. Epub 2007 Jun 28. PMID 17655972
- [Derived] Hollingworth S, Dalton M, Blundell JE, Finlayson G. Evaluation of the Influence of Raw Almonds on Appetite Control: Satiation, Satiety, Hedonics and Consumer Perceptions. Nutrients. 2019 Aug 30;11(9):2030. doi: 10.3390/nu11092030. PMID 31480245

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Start Date: June 2015
  Recruitment End Date: October 2015
  Responses to Study Advertisement: 303
  Number of Participants Invited to Screening Session: 85
  Number of Participants Screened: 49
  Number of Participants Recruited: 42
  Number of Participants Completed: 42
Groups:
- Almond, Then No Food, Then Cheese Savouries: Participants first received a mid-morning snack of almonds. After a washout period of 5 days, they then received no food. Finally, after another washout period participants received a mid-morning snack of cheese savouries.
- Cheese Savouries Then Almond, Then No Food: Participants first received a mid-morning snack of cheese savouries. After a washout period of 5 days, they then received a mid-morning snack of almonds. Finally, after another washout period participants received no food.
- No Food, Then Cheese Savouries, Then Almond: Participants first received no food. After a washout period of 5 days, they then received a mid-morning snack of cheese savouries. Finally, after another washout period participants received a mid-morning snack of almonds.
- Cheese Savouries, Then No Food, Then Almond: Participants first received a mid-morning snack of cheese savouries. After a washout period of 5 days, they then received no food. Finally, after another washout period participants received a mid-morning snack of almonds.
- Almond, Then Cheese Savouries, Then No Food: Participants first received a mid-morning snack of almonds. After a washout period of 5 days, they then received a mid-morning snack of cheese savouries. Finally, after another washout period participants received no food.
- No Food, Then Almond, Then Cheese Savouries: Participants first received no food. After a washout period of 5 days, they then received a mid-morning snack of almonds. Finally, after another washout period participants received a mid-morning snack of cheese savouries.
Period: Overall Study
Arm/Group | Almond, Then No Food, Then Cheese Savouries | Cheese Savouries Then Almond, Then No Food | No Food, Then Cheese Savouries, Then Almond | Cheese Savouries, Then No Food, Then Almond | Almond, Then Cheese Savouries, Then No Food | No Food, Then Almond, Then Cheese Savouries
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed all three study conditions were included in the analyses.
Groups:
- Overall Sample: Dosage was 0.9g/kg of 1) Whole raw almonds, 2) Cheese savoury crackers, 3) no food given in a randomised cross-over design with order determined by Latin square (i.e. 6 order permutations). Doses were administered once as a mid-morning snack.
Arm/Group | Overall Sample
Number analyzed (Participants) | 42
Age, Continuous [Median (Standard Deviation); unit: Years] | 26.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Weight [Mean (Standard Deviation); unit: kg] | 58.5 (6.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.0 (2.0)
Waist [Mean (Standard Deviation); unit: cm] | 73.5 (5.6)
Fat Mass [Mean (Standard Deviation); unit: kg] | 15.4 (5.0)
Fat Free Mass [Mean (Standard Deviation); unit: kg] | 43.0 (4.1)
Body Fat Percentage [Mean (Standard Deviation); unit: %] | 26.0 (6.7)
Three Factor Eating Questionnaire - Restraint subscale [Mean (Standard Deviation); unit: units on a scale] — Cognitive restraint over eating. Scale range: 0-21 Higher values indicate greater restraint over eating
  units on a scale | 9.4 (4.8)
Three Factor Eating Questionnaire - Disinhibition subscale [Mean (Standard Deviation); unit: units on a scale] — Disinhibition of restraint Scale range: 0-16 Higher scores indicate worse outcome
  units on a scale | 7.6 (2.8)
Three factor Eating Questionnaire - Hunger subscale [Mean (Standard Deviation); unit: units on a scale] — Susceptibility to hunger Scale range: 0-13 Higher scores indicate worse outcome
  units on a scale | 6.1 (3.2)
Binge Eating Scale [Mean (Standard Deviation); unit: units on a scale] — Binge eating scale Scale range: 0-46 Higher scores indicate worse outcome
  units on a scale | 10.1 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Test Meal Energy Intake
Description: Measured reductions in ad-libitum energy intake following consumption of almonds as a mid-morning snack compared to control and comparator. Food will be weighed pre- and post-consumption to the nearest 0.1g to determine energy intake. Test meal energy intake will be measured on three occasions, on average a week apart.
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: kcal
Groups:
- Almonds: Whole, raw almonds Almonds
- Cheese Savouries: Sainsbury's savoury biscuits Cheese Savouries
- No Food: No food provided, just water
Arm/Group | Almonds | Cheese Savouries | No Food
Number analyzed (Participants) | 42 | 42 | 42
kcal | 1007.3 (299.1) | 1019.6 (345.6) | 1143.4 (347.4)
Statistical Analysis 1: Comparison: Almonds vs Cheese Savouries vs No Food; Test type: Superiority or Other; p < 0.01, ANOVA — Where significant effects were obtained post hoc analyses, with a Bonferroni correction for multiple comparisons were conducted; Null hypothesis is that there was no difference in energy intake between almonds, cheese savouries and no food

2. Secondary Outcome: Food Preference
Description: Measured changes in wanting for high fat food food following consumption of almonds as a mid-morning snack compared to control and comparator.
  Food preference will be measured once during each intervention condition using the Leeds Food Preference Questionnaire (LFPQ: Finlayson, King & Blundell, 2008).
  8 high fat foods and 8 low fat foods are presented on a computer and participants rate the extent to which they want each food (How much do you want this food now?). The food images are presented individually, in a randomised order and participants make their ratings using a 100-mm VAS. Low fat scores are subtracted from high fat scores to provide a relative preference score.
  Scale range: -100 to 100. Higher scores indicate greater wanting for high fat foods which is interpreted as a worse outcome.
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Almonds | Cheese Savouries | No Food
Number analyzed (Participants) | 42 | 42 | 42
units on a scale | 10.56 (30.6) | 5.45 (40.1) | 20.30 (27.7)
Statistical Analysis 1: Comparison: Almonds vs Cheese Savouries vs No Food; Test type: Superiority or Other; p < 0.05, ANOVA — [p-value comment as in outcome 1, analysis 1]; Null hypothesis is that there was no difference in wanting for high fat foods between almonds, cheese savouries and no food

3. Secondary Outcome: Appetite Sensations (Hunger)
Description: Measured differences in hunger following consumption of almonds as a mid-morning snack compared to control and comparator.
  Appetite sensations will be measured during the three intervention conditions at regular time intervals from the morning to the evening (21 in total) using 100-mm visual analogue scale (VAS).
  Scale range = 0-100 mm, with higher values indicating greater hunger. Total Area Under the Curve will be calculated from the VAS profiles using the trapeziodal method.
  Time points at which data were collected to calculate AUC - -5, 15, 30, 60, 90, 120, 135, 180, 230, 240, 270, 280, 300, 360, 420, 480, 510, 540, 600; -5 to 8 hours post intervention.
  Higher AUC scores on hunger are interpreted as a worse outcome.
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: minutues*mm
Arm/Group | Almonds | Cheese Savouries | No Food
Number analyzed (Participants) | 42 | 42 | 42
minutues*mm | 11207.2 (5915.9) | 13328.0 (6342.6) | 14638.4 (5288.2)
Statistical Analysis 1: Comparison: Almonds vs Cheese Savouries vs No Food; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Null hypothesis is that there was no difference in hunger AUC between almonds, cheese savouries and no food

4. Secondary Outcome: 24 Hour Energy Intake
Description: Measured reductions in total within-day energy intake following consumption of almonds as a mid-morning snack compared to control and comparator. Food will be weighed pre- and post-consumption to the nearest 0.1g, at every test meal, to determine energy intake. Total energy intake will then be calculated. 24 hour energy intake will be measured on three occasions, on average a week apart.
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Almonds | Cheese Savouries | No Food
Number analyzed (Participants) | 42 | 42 | 42
kcal | 2992.0 (654.2) | 2990.6 (748.9) | 2797.2 (728.2)
Statistical Analysis 1: Comparison: Almonds vs Cheese Savouries vs No Food; Energy intake measured by ad-libitum test meals (breakfast, lunch, dinner) during each intervention condition. Null hypothesis is that there was no difference in total energy intake between almonds, cheese savouries and no food; Test type: Superiority or Other; p < 0.05, ANOVA; Null hypothesis is that there was no difference in energy intake between almonds, cheese savouries and no food

ADVERSE EVENTS:
Time Frame: 6 months (June 15 - November 15)
Groups:
- Almond, Then No Food, Then Cheese Savouries: Participants first received a mid-morning snack of almonds. After a washout period of 5 days, they then received no food. Finally, after another washout period participants received a mid-morning snack of cheese savouries.
  Dosage was 0.9g/kg of 1) Whole raw almonds, 2) Cheese savoury crackers, 3) no food given in a randomised cross-over design with order determined by Latin square (i.e. 6 order permutations). Doses were administered once as a mid-morning snack.
- Cheese Savouries Then Almond, Then No Food: Participants first received a mid-morning snack of cheese savouries. After a washout period of 5 days, they then received a mid-morning snack of almonds. Finally, after another washout period participants received no food.
  Dosage was 0.9g/kg of 1) Whole raw almonds, 2) Cheese savoury crackers, 3) no food given in a randomised cross-over design with order determined by Latin square (i.e. 6 order permutations). Doses were administered once as a mid-morning snack.
- No Food, Then Cheese Savouries, Then Almond: Participants first received no food. After a washout period of 5 days, they then received a mid-morning snack of cheese savouries. Finally, after another washout period participants received a mid-morning snack of almonds.
  Dosage was 0.9g/kg of 1) Whole raw almonds, 2) Cheese savoury crackers, 3) no food given in a randomised cross-over design with order determined by Latin square (i.e. 6 order permutations). Doses were administered once as a mid-morning snack.
- Cheese Savouries, Then No Food, Then Almond: Participants first received a mid-morning snack of cheese savouries. After a washout period of 5 days, they then received no food. Finally, after another washout period participants received a mid-morning snack of almonds.
  Dosage was 0.9g/kg of 1) Whole raw almonds, 2) Cheese savoury crackers, 3) no food given in a randomised cross-over design with order determined by Latin square (i.e. 6 order permutations). Doses were administered once as a mid-morning snack.
- Almond, Then Cheese Savouries, Then No Food: Participants first received a mid-morning snack of almonds. After a washout period of 5 days, they then received a mid-morning snack of cheese savouries. Finally, after another washout period participants received no food.
  Dosage was 0.9g/kg of 1) Whole raw almonds, 2) Cheese savoury crackers, 3) no food given in a randomised cross-over design with order determined by Latin square (i.e. 6 order permutations). Doses were administered once as a mid-morning snack.
- No Food, Then Almond, Then Cheese Savouries: Participants first received no food. After a washout period of 5 days, they then received a mid-morning snack of almonds. Finally, after another washout period participants received a mid-morning snack of cheese savouries.
  Dosage was 0.9g/kg of 1) Whole raw almonds, 2) Cheese savoury crackers, 3) no food given in a randomised cross-over design with order determined by Latin square (i.e. 6 order permutations). Doses were administered once as a mid-morning snack.
Arm/Group | Almond, Then No Food, Then Cheese Savouries | Cheese Savouries Then Almond, Then No Food | No Food, Then Cheese Savouries, Then Almond | Cheese Savouries, Then No Food, Then Almond | Almond, Then Cheese Savouries, Then No Food | No Food, Then Almond, Then Cheese Savouries
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/7 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No